CLINICAL TRIAL: NCT04600622
Title: Adapting and Assessing the Feasibility of a Diabetes Self-management Education and Support Telehealth Intervention for Rural Populations to Reduce Disparities in Diabetes Care
Brief Title: Adapting and Assessing the Feasibility of a Diabetes Self-management Telehealth Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Michelle Litchman, Assistant Profesor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00133179
Record Dates: First submitted 2020-10-15; First posted 2020-10-23 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; telehealth; rural; Spanish; English; community based participatory research
MeSH Terms: conditions — Diabetes Mellitus | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants will receive Rural Diabetes One-Day Education and Care program (R-D1D). A one time, 5.5-hour multi-disciplinary diabetes self-management education and support intervention delivered via telehealth.
  Interventions: Behavioral: Rural Diabetes One-Day Education and Care program (R-D1D)
- Active Comparator (Active Comparator): Participants will receive diabetes education materials.
  Interventions: Behavioral: Diabetes Education Materials

INTERVENTIONS:
Behavioral: Rural Diabetes One-Day Education and Care program (R-D1D) — One time, 5.5-hour multi-disciplinary diabetes self-management education and support intervention delivered via telehealth.
  Arms: Intervention Arm
Behavioral: Diabetes Education Materials — Diabetes Education Materials
  Arms: Active Comparator

SUMMARY:
The proposed project will use community based participatory research to adapt an existing diabetes self-management and education intervention with a telehealth intervention to be culturally relevant for rural English- and Spanish-speaking populations. Participants and care partners will receive a one-time, 5.5-hour telehealth intervention from a multidisciplinary team specializing in diabetes. The overarching aim of this study is to provide a sustainable model to provide diabetes specialty care to rural populations.

DETAILED DESCRIPTION:
Diabetes prevalence is higher in rural areas that have lower resources to diabetes self-management education and support (DSMES), a cornerstone to optimal diabetes management. A time efficient DSMES program delivered via telehealth by multidisciplinary experts that also encourages care partner and peer support is a creative solution to increasing access to DSMES and reducing disparities. This study is guided by the Research, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework. English and Spanish-speaking participants and care partners will receive a one-time, 8-hour telehealth intervention at the rural clinic where they receive their usual care, from the multidisciplinary team. The rural clinical practices will provide feedback in two rounds, with iterative practice-level changes, to address process and/or workflow issues. Our overall objective is to adapt, implement, refine, and evaluate a time efficient DSMES program delivered via telehealth by a team of multidisciplinary experts that encourages care partner and peer support to improve A1C and diabetes self-management in rural communities to reduce disparities. Our multidisciplinary team includes researchers and clinical healthcare providers with experience in diabetes care, DSMES delivery, community-engaged research, practice-based research, and rural health issues. The University of Utah and High Plains Research Network provide a strong environment for this particular study. The proposed study will 1) adapt the exiting Diabetes One-Day Program (D1D) for use in rural communities (Rural Diabetes One-Day Program or R-D1D), 2) conduct a patient-level pilot RCT to examine effects of R-D1D (intervention group) versus standard patient education (attention control group), guided by the RE-AIM framework. Our ultimate goal is to reduce health disparities in rural populations by increasing access to diabetes specialty care using telehealth. Preliminary data support the D1D intervention, but will require adaptation to translate for rural populations, then iterative refinement at the practice level to support long-term maintenance. Such a tested, accepted intervention should have a beneficial effect on diabetes self-management across multiple rural locations.

ELIGIBILITY:
Inclusion Criteria:

* Have a known diagnosis of type 1 or 2 diabetes with any A1C level
* 18 years old or older
* Live in a rural eastern Colorado
* Speak and understand English or Spanish
* Willing to participate in a telehealth intervention at the clinic where they usually receive care or in their own home if an in-person meeting is prohibited due to the pandemic

Exclusion Criteria:

* Are participating in another diabetes study
* Significant cognitive impairment
* Pregnant or planning to become pregnant as diabetes management recommendations are different in pregnancy
* Life expectancy of <6 months
* Plan to move during the time of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Average Acceptability Score | 3 months
  Average acceptability score on the intervention acceptability measure
Average Feasibility Score | 3 months
  Average feasibility score on the feasibility measure

SECONDARY OUTCOMES:
Change in glycosylated hemoglobin A1C | Baseline to 3 months
  Physiologic measurement
Change in diabetes distress score | Baseline to 3 months
  The patient reported, 20-item, Problem Areas in Diabetes survey will be used.
Change in Family and Friend Involvement in Diabetes score | Baseline to 3 months
  The patient reported, 16-item, Family and Friend Involvement in Diabetes survey will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L Litchman, PhD, Principal Investigator — University of Utah College of Nursing; Tamara K Oser, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Litchman ML, Kwan BM, Zittleman L, Simonetti J, Iacob E, Curcija K, Neuberger J, Latendress G, Oser TK. A Telehealth Diabetes Intervention for Rural Populations: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Jun 14;11(6):e34255. doi: 10.2196/34255. PMID 35700026